CLINICAL TRIAL: NCT04804826
Title: Patient's Perceptions Regarding Same Day Discharge Following Pelvic Reconstructive Surgery: What do They Want Other Patients to Know?
Brief Title: Same Day Discharge Following Pelvic Reconstructive Surgery
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 21-010
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Same Day Discharge; Pelvic Organ Prolapse; Total Vaginal Hysterectomy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pelvic Reconstructive Surgery — Pelvic Reconstructive Surgery including total vaginal hysterectomy

SUMMARY:
This is a prospective cross-sectional study in which patients undergoing major pelvic reconstructive surgery with total vaginal hysterectomy will be recruited and enrolled. At approximately 2 weeks and 12 weeks postoperatively, enrolled patients will be asked to complete a survey detailing their experience with SDD, surgical recovery, and advice for prospective patients.

ELIGIBILITY:
Inclusion Criteria:

* Total vaginal hysterectomy with or without bilateral salpingectomy/oophorectomy
* Apical repair with uterosacral ligament suspension or sacrospinous ligament fixation
* They may also have any of the following concurrent procedures: Anterior repair, Posterior repair, Enterocele repair, Suburethral sling for incontinence
* Surgery by one of the fellowship trained urogynecologists at TriHealth
* English speaking

Exclusion Criteria:

* Enrollment in the "Diazepam Research Study" (Protocol ID:19-130)
* Concomitant procedure with another surgeon
* Chronic pain conditions that require daily use of narcotic pain medications (including but not limited to: chronic back or pelvic pain, interstitial cystitis, fibromyalgia)
* Concomitant anal sphincteroplasty, mesh removal or use of mesh for prolapse (excluding sling procedures)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent a total vaginal hysterectomy with concurrent vaginal native tissue prolapse repairs, including an apical suspension procedure performed by one of the fellowship trained urogynecologists at TriHealth.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Number of subjects who satisfied with the results of the surgery | Approximately 2 weeks postoperatively
  Number of subjects who answered either "Very Satisfied" or "Satisfied" to a Likert scale question "How satisfied are you with the results of your surgery." The liker scale choices are "Very Satisfied", "Satisfied", "Neutral", "Unsatisfied", and "Very Unsatisfied."

SECONDARY OUTCOMES:
Number of subjects who satisfied with the results of the surgery | Approximately 12 weeks postoperatively
  Number of subjects who answered either "Very Satisfied" or "Satisfied" to a Likert scale question "How satisfied are you with the results of your surgery." The liker scale choices are "Very Satisfied", "Satisfied", "Neutral", "Unsatisfied", and "Very Unsatisfied."

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Lloyd JC, Guzman-Negron J, Goldman HB. Feasibility of same day discharge after robotic assisted pelvic floor reconstruction. Can J Urol. 2018 Jun;25(3):9307-9312. PMID 29900817
- [Background] Evans S, Myers EM, Vilasagar S. Patient perceptions of same-day discharge after minimally invasive gynecologic and pelvic reconstructive surgery. Am J Obstet Gynecol. 2019 Dec;221(6):621.e1-621.e7. doi: 10.1016/j.ajog.2019.06.046. Epub 2019 Jun 27. PMID 31254524